CLINICAL TRIAL: NCT01248676
Title: An Evaluation of the Usability and Usefulness of a Multi-language Online Patient Education Module: A Pilot Study
Brief Title: An Evaluation of the Usability and Usefulness of a Multi-language Online Patient Education Module
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Lisa Di Prospero, Odette Cancer Centre at Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Cindy Multi-Language Online
Record Dates: First submitted 2010-11-18; First posted 2010-11-25 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Cancer
Keywords: cancer radiation patient education
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Multi-language Online Patient Education Module in addition to standard Patient Teaching — Patients are usually be given a 5-10 minute "new patient teaching" before their radiation therapy simulation and planning appointment and before their first radiation therapy treatment appointment. Patients will be asked to view an online patient education module before their radiation therapy simulation and planning appointment or before their first radiation therapy treatment appointment. Then patients will be asked to participate in an interview session and fill out a survey (attached). They will still receive "new patient teaching" from the therapists before their radiation therapy simulation and planning or radiation therapy treatment appointment.

SUMMARY:
The purpose of this study is to determine if multi-language patients will find the multi-language capabilities of the online modules useful for better understanding of the general information regarding radiation therapy.

DETAILED DESCRIPTION:
Research shows that treatment-related information is the most important informational need of cancer patients and online media sources are gaining popularity as a cancer communication method. It is important to know whether having multi-language online education modules are usable for and beneficial to the multicultural cancer patient population at Sunnybrook Hospital, given that recent research suggests that this cancer population in general faces many barriers to effective online cancer communication. Approximately 10 new patients from the radiation oncology clinic at Sunnybrook Hospital will be screened to participate in the study. Usability testing will involve a combination of interviewing, observation, think-aloud methodology and a short survey.Results will be analyzed by assessing the percentage of patients identifying with a certain level of the Likert scale on the survey as well as through content analysis of responses to the interview and open-ended survey questions.

ELIGIBILITY:
Inclusion Criteria:

* first/second language in one of the module languages with the ability to understand and communicate English to an understandable degree, basic computer skills, and the ability to complete 20-30 minutes of testing.

Exclusion Criteria:

* inability to participate in 20-30 minutes of usability testing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Patients will be asked to give their rating (Likert scale) on the usefulness of the information on the patient education site with regard to their upcoming radiation simulation and treatment. | Within one month of patients initial consultation with the Radiation Oncologist

SECONDARY OUTCOMES:
Patients will be asked to give their rating (Likert scale) on how easily the online patient education module is to navigate. | Within one month of patients initial consultation with the Radiation Oncologist

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S Di Prospero, MSc, Principal Investigator — Odette Cancer Centre at Sunnybrook Health Sciences Centre
Locations (1):
- Odette Cancer Centre at Sunnybrook Health Sciences, Toronto, Ontario, Canada